CLINICAL TRIAL: NCT05482425
Title: A Single Center, Randomized Study to Evaluate Skin Characteristics After Facial Autologous Fat Grafting to Both Sides of the Face Using Saline Washed or Unwashed Fat Graft.
Brief Title: Autologous Facial Fat Grafting Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, J. Peter Rubin, MD, UPMC Endowed Professor and Chair of Plastic Surgery, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY21110089
Record Dates: First submitted 2022-03-16; First posted 2022-08-01 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-11

CONDITIONS: Facial Skin Texture; Facial Skin Pigmentation

STUDY DESIGN:
Intervention Model Description: This study will include 2 cohorts, each consisting of approximately 13 subjects to undergo intervention, where each subject will have treatment of the skin of cheek area, upper lip, chin and superior neck regions, as well as the behind the ears with autologous fat graft. The subject will receive either a saline washed preparation or a non-washed preparation as determined by the randomization process. Autologous fat tissue will be harvested for the fat graft preparation (up to a maximum of 1 liter ) from the trunk or extremity donor site, consistent with standard clinical practice.
Who Masked: Outcomes Assessor
Masking Description: Blinded grading based on VECTRA images and VISIA images will be performed on de-identified photography by a third-party vendor at the end of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Autologous facial fat graft injection- washed fat (Other): Washed fat injected into both the left and right sides of the face.
  Interventions: Other: Autologous facial fat graft injection
- Autologous facial fat graft injection-unwashed fat (Other): Unwashed fat injected into both the left and right sides of the face.
  Interventions: Other: Autologous facial fat graft injection

INTERVENTIONS:
Other: Autologous facial fat graft injection — Participants will received either a washed or unwashed autologous facial fat graft injection to both sides of the face, as determined by randomization.

SUMMARY:
The goal of this study is to specifically examine changes in facial skin appearance after facial fat grafting with autologous fat tissue that has either been washed with sterile saline before injecting, or left unwashed. This will be testing two variations of a standard of care surgical procedure, in two cohorts of subjects. One group will receive washed fat, and one group will receive unwashed fat, to both sides of the face. There are no experimental devices, drugs, or biological agents being used in this study. All fat tissue is autologous from the subjects treated.

Significance: This study will provide evidence that may directly impact clinical practice for a common procedure in plastic surgery. Regardless of whether the null hypotheses is accepted or rejected, the data will be of direct clinical use and impact practice in the operating room.

DETAILED DESCRIPTION:
Autologous fat grafting is a very common standard of care procedure in plastic surgery, used for both aesthetic and reconstructive applications across the entire body.1 Facial fat grafting, in particular, is the most common site for use of autologous fat. The American Society of Plastic Surgeons (ASPS) statistics report showed 133,720 cases of facial fat grafting for cosmetic indications in 2020.2 This is mainly due to the fact that humans lose facial fat during the aging process, and that loss of volume leads to characteristic signs of aging.3 It is also well known that when autologous fat grafting is used for facial cosmetic injections, increasing the amount of fat in the dermal/subdermal region has very positive effects on the appearance of the skin.4-6 This is because adding more padding beneath the skin gives the appearance of suppleness and smoothness and mitigates the "deflated" appearance that patients complain of. Additionally, as the adipose graft tissue heals, it tends to increase vascularization in the region which also has a positive effect on the skin. This can improve fine and course wrinkles, and color tone and pigmentary variation can also improve.7-9 Facial fat grafting is commonly performed by surgeons at UPMC and throughout the Pittsburgh region, consistent with national practice patterns.

Autologous fat grafting is a minimally invasive procedure that involves harvest of fat tissue with a liposuction cannula. In many cases, the cannula is attached to a 10 mL syringe and negative pressure applied by withdrawing the syringe plunger during aspiration.1 In other cases, a mechanical aspiration machine is used to generate negative pressure.1 Either way, all of this equipment is standard in most operating rooms across the country. The aspirated material consists of small particles of adipose tissue, measuring between three and five mm in diameter.10 Once harvested into sterile vessels, the aspirate can be gently centrifuged or strained to separate and remove the aqueous and oil layers. If washed, a sterile saline solution would be used to perform the washing procedure. The material is often transferred between syringes using a Luer Lock connector and the graft material is then injected from syringes. Passing the tissue multiple times between Luer Lock connectors has become a very common method of breaking up clumps of tissue and enabling a more flowable graft material that can be injected through smaller gauge cannula without clogging.11

Controversy exists in the plastic surgery community as to the most beneficial preparation methods in the operating room.12 Different surgeons use a number of methods alone or in combination that include filtering or straining fat, gentle centrifugation, separation of fluid and oil layers by gravity, and rinsing/washing with sterile saline. All of these methods are well accepted as within standard of care and represent minimal manipulation of the tissue grafts. A national survey of the plastic surgery community, published by our group revealed that 28% of surgeons use a saline wash during their fat graft processing.13 The rationale for a saline wash is that it may decrease any residual free lipid/oil, as well as residual red cells, both of which can potentially cause irritation of the local tissues. However, opponents of washing often cite that there washing adds an extra step without clinical benefit.

Hypothesis: We hypothesize that a saline washed fat graft injectate will have improved appearance of facial skin. We speculate that the reduced free lipid and reduced red cell fraction will be beneficial in the healing process.

Significance: This study will provide evidence that may directly impact clinical practice for a common procedure in plastic surgery. Regardless of whether the null hypotheses is accepted or rejected, the data will be of direct clinical use and impact practice in the operating room.

Treatment Period: Autologous fat graft injections will be performed on Day 0 of the study period after eligibility determination has been made, and after baseline data collection. Subjects will be followed over a 12-month time period.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to perform informed consent
2. Healthy female adults, from 35 to 70 years of age
3. Fitzpatrick Skin Type Scale scores < 3.
4. FWAS-greater than moderate, equal to or greater than 4
5. Noticeable Physical signs of facial aging and sun damage including skin wrinkles, loss of elasticity and pigmentary changes, with greater than mild (≥4 on a 0 to 9 scale) signs of the following, per investigator discretion

   1. Facial wrinkles (periorbital//periorbital//cheek)
   2. Dyschromia (hyperpigmentation//uneven skin tone)
   3. Rough skin texture (visual skin roughness//pore sizes)
6. Willingness to undergo the proposed treatment and comply with study procedures.
7. Negative pregnancy urine dip test (as indicated-unless s/p hysterectomy or past menopause documentation can be sourced to research chart.)
8. Willingness to avoid the use of laser, IPL, Botox (6 months), injectable fillers or other surgical cosmetic procedures on the face for 6 months ducts
9. Ability to produce sufficient fat tissue from donor site during harvest (up to a maximum of 1 liter)

Exclusion Criteria:

1. Age < 35 or > 70 years of age
2. Any medical condition that would preclude safe administration of anesthesia and safe conduct of the adipose harvest procedure (such as an uncontrolled bleeding disorder or severe pulmonary disease), per investigator discretion.
3. Active infection on the face (e.g., acne, HSV (herpes simplex), etc.,) per investigator discretion.
4. Female in pregnancy (positive pregnancy-test performed before inclusion) or lactation or without effective contraception)
5. Received laser, IPL, botox (6 months), injectable fillers or other surgical cosmetic procedures on the face within 12 months of study consent and screening date. -prohibited for 6 months
6. Acutane use within past 12 months
7. Individuals with any contraindications of autologous lipografting, such as cutaneous rashes or infection in the area of intended fat harvest, lack of available donor fat, or other factors that, in the determination of the investigator, would be considered a contraindication.
8. Individuals diagnosed with known allergies to skin care products, topical antibiotics, adhesives, bandages, lidocaine, epinephrine, or other agents that might be used in the study
9. Individuals with any disease state or inappropriate physical skin condition (e.g., active/history of psoriasis, active eczema, excessive hair, scars, tattoos, etc. on face) that might impair evaluations or increase the health risk to the subject by participation in the opinion of the Investigator
10. Individuals with a history of immunosuppression/immune deficiency disorders/ known or suspected defect of healing (including HIV infection or AIDS)
11. Individuals with an uncontrolled disease such as hypertension, hyperthyroidism, or hypothyroidism, which may impact safety. Individuals having multiple health conditions may be excluded from participation even if the conditions are controlled by diet, medication, which in the opinion of the Investigator, may create safety concerns or interfere with the study.
12. Individuals currently taking substances known to affect bleeding time, which in the opinion of the Investigator, may create safety concerns or interfere with the study (e.g., aspirin, Heparin, Warfarin, Plavix, supplements, etc.).
13. Individuals currently and chronically taking substances known to impair the immune system at doses anticipate to have a systemic effect on wound healing (e.g., corticosteroids, immunosuppressant, etc. or currently using immunosuppressive medications (e.g., azathioprine, belimumab, cyclophosphamide, Enbrel, Imuran, Humira, mycophenolate mofetil, methotrexate, prednisone, Remicade, Stelara.) within 30 days of the study start and in the discretion of the PI would impact the results of the study. Steroid treatments that would not be expected to impact study results could include steroid inhaler, nasal spray, eyedrops, topical creams used in areas outside of the face, or transient oral dose of steroids to treat acute conditions (eg pulsed oral dose for respiratory airway constriction or skin rash)
14. Individuals with a history of documented keloid scar formation, prominent skin lesions or scars that would render data collection and aesthetic evaluation impossible. The investigator will make that determination based on examining other scars and reviewing any history of treatment for keloid lesions.
15. Individuals with a diagnosis of diabetes
16. Subject participating in another interventional clinical trial assessing treatments that may interfere with the accuracy of data collection for this study within 1 month of Visit 1
17. The inability to obtain sufficient fat from the donor site during the harvest to allow the autologous fat tissue processing prior to facial injection.

Ages: 35 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Healthy female adults, from 35-70 years of age
Enrollment: 26 (Actual)
Dates: Start 2022-10-17 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Change in facial skin characteristics as measured by the Fitzpatrick Wrinkle Scale (FWAS) from baseline to 12 month assessment, compared between the two cohorts. Scale (FWAS) from baseline to 12 month assessment, compared between the two cohorts. | Baseline, 12 months
  The Fitzpatrick Wrinkle Assessment (FWAS); The FWAS quantifies the degree of wrinkling and elastosis in subjects on a scale of 0 to 9, zero being the best possible condition and 9 to be considered the worst possible condition. Change from baseline within each subject will be calculated from baseline up to 12 month using the FWAS Score, and then overall changes compared between the two cohorts.
Change in facial skin characteristics as measured by the Skin Quality Assessment (SQA) form from baseline up to 12 month assessment, compared between the two cohorts. | Baseline, 12 months
  Skin Quality Assessment (SQA): The SQA assesses skin quality scale in terms of four categories: tone (dyschromia), elasticity (firmness), texture (smoothness), and radiance (brightness). Each of these four categories are measured on a scale of 0 to 4, with 0 being the best possible condition and 4 being the worst possible condition Change from the baseline within each subject will be calculated using the SQA score from baseline up to 12 month, and then overall changes compared between the two cohorts.
Change in facial skin characteristics as measured by the Subject Satisfaction Scale (SSA) form from baseline up to 12 month assessment, compared between the two cohorts. | Baseline, 12 months
  Subject Satisfaction Scale (SSA):The SSA was designed to assess subject overall satisfaction with rejuvenation treatment and skin care products. The scale is defined as following:
  * 3 (very dissatisfied)
  * 2 (dissatisfied)
  * 1 (somewhat dissatisfied) 0 (neutral)
    1. (somewhat satisfied)
    2. (satisfied)
    3. (very satisfied) Change from baseline within each subject will be calculated using the SSA score from baseline up to 12 month, and then overall changes compared between the two cohorts.
Self esteem as measured by the Heatherton and Polivy State Self Esteem Scale (SESS) form from baseline to 12 month assessment, compared between the two cohorts. | Baseline, 12 months
  Heatherton and Polivy State Self-Esteem Scale (SESS); The SSES is a validated instrument with multiple statements characterizing self-esteem on a scale from one to 5. (One being no self-esteem and five being extreme self-esteem.) Change from baseline within each subject will be calculated using the SESS score from baseline to 12 month, and then overall changes compared between the two cohorts.
Change in facial skin characteristics as measured by the Global Aesthetic Improvement Scale (GAIS) form from baseline to 12 month assessment, compared between the two cohorts. | Baseline, 12 months
  Global Aesthetic Improvement Scale (GAIS); The GAIS is a validated five-point relative improvement scale. This scale has been used in previous studies to evaluate for change in subject appearance following treatment. The scale is defined as following:
  1. Exceptional improvement
  2. Very improved patient
  3. Improved patient
  4. Unaltered patient
  5. Worsened patient
  Change from baseline within each subject will be calculated using the GAIS score from baseline to 12 month, and then overall changes compared between the two cohorts.
Change in facial skin characteristics as measured by the Participant Satisfaction questionnaire from baseline to 12 months, compared between the two cohorts. | 12 month
  Participant Satisfaction Questionnaire- participants will be asked to rate their facial appearance in specific aspects of the face such as cheek wrinkles, skin clarity, and skin smoothness, etc., using a 9 point scale (with 0 being the best possible condition and 9 being the worst possible condition. In addition, participants will rate level of their perceived level of improvement in those same facial aspects on a 9 point scale,. Change within each subject will be calculated using the participant satisfaction questionnaire score from baseline to 12 month, and then overall rates compared between the two cohorts.
Change in facial skin characteristics as measured by the cutometer from baseline up to 12 months, compared between groups. | Baseline, 12 months
  Assessment of skin elasticity by Cutometer® Dual MPA 580: The instrument applies a vacuum to a small area of skin, and measures the elastic response of the skin. The probe will be kept at a 90# angle during the measurements. This assessment will be performed on each side of the face at the intersection of lines extending down from the center of the eye and horizontally across the bottom of the nose. Reduction in wrinkle size will be assessed at baseline and 12 months, and overall rate of change compared between the two cohorts.

SECONDARY OUTCOMES:
Change in facial skin characteristics by expert graders using a Griffth scale. | Baseline, 12 months
  Facial skin characteristics such as including Crow's feet area wrinkles, under eye area wrinkles, perioral wrinkles, skin tone evenness, skin pigmentation, skin texture, skin radiance and overall skin health will be rated using the Griffth scale. The Griffth scale is scored on a 0 to 9 scale with 0 being the best possible condition and 9 being the worst possible condition, based on 2D and 3D images captured during the study. Change from baseline within each subject will be calculated from baseline up to 12 months using the Griffth's scale, and then overall changes compared between the two cohorts.
Compare investigator's rating of the change in facial skin characteristics, as recorded during baseline and 12 month history and physical exam form, compared between the two cohorts. | Baseline, 12 months
  The investigator will record on the History and Physical exam form whether skin characteristics such as facial wrinkles (crow's feet, cheek), hyperpigmentation, uneven skin tone, skin roughness and pore size are present at baseline. At the follow up 12 month visit, the investigator will record whether these characteristics have improved since baseline (Yes/No). Rates of improvement will be calculated within each cohort and then compared between the two groups.
To assess the safety of the autologous fat injections, compared between the two cohorts, from baseline to 12 months. | Baseline, 12 months
  Number of participants with at least one adverse event will be counted, AEs will be summed per cohort, and rates compared between the two groups.

CONTACTS AND LOCATIONS:
Overall Officials: J. Peter Rubin, MD, Principal Investigator — University of Pittsburgh; Patsy Simon, BS, RN, CCRC, CCRA, ACRP-PM, Study Director — University of Pittsburgh
Locations (1):
- UPMC Aesthetic Plastic Surgery Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Strong AL, Cederna PS, Rubin JP, Coleman SR, Levi B. The Current State of Fat Grafting: A Review of Harvesting, Processing, and Injection Techniques. Plast Reconstr Surg. 2015 Oct;136(4):897-912. doi: 10.1097/PRS.0000000000001590. PMID 26086386
- [Background] Plastic Surgery Statistics. Plastic surgery procedural statistics from the American Society of Plastic Surgeons. Accessed January 21, 2022. https://www.plasticsurgery.org/news/plastic-surgery-statistics
- [Background] Wollina U, Wetzker R, Abdel-Naser MB, Kruglikov IL. Role of adipose tissue in facial aging. Clin Interv Aging. 2017 Dec 6;12:2069-2076. doi: 10.2147/CIA.S151599. eCollection 2017. PMID 29255352
- [Background] Egro FM, Coleman SR. Facial Fat Grafting: The Past, Present, and Future. Clin Plast Surg. 2020 Jan;47(1):1-6. doi: 10.1016/j.cps.2019.08.004. Epub 2019 Oct 21. PMID 31739886
- [Background] Schultz KP, Raghuram A, Davis MJ, Abu-Ghname A, Chamata E, Rohrich RJ. Fat Grafting for Facial Rejuvenation. Semin Plast Surg. 2020 Feb;34(1):30-37. doi: 10.1055/s-0039-3402767. Epub 2020 Feb 15. PMID 32071577
- [Background] Marten T, Elyassnia D. Facial Fat Grafting: Why, Where, How, and How Much. Aesthetic Plast Surg. 2018 Oct;42(5):1278-1297. doi: 10.1007/s00266-018-1179-x. Epub 2018 Aug 31. PMID 30171292
- [Background] Coleman SR. Structural fat grafting: more than a permanent filler. Plast Reconstr Surg. 2006 Sep;118(3 Suppl):108S-120S. doi: 10.1097/01.prs.0000234610.81672.e7. PMID 16936550
- [Background] Evans BGA, Gronet EM, Saint-Cyr MH. How Fat Grafting Works. Plast Reconstr Surg Glob Open. 2020 Jul 14;8(7):e2705. doi: 10.1097/GOX.0000000000002705. eCollection 2020 Jul. PMID 32802628
- [Background] Mojallal A, Lequeux C, Shipkov C, Breton P, Foyatier JL, Braye F, Damour O. Improvement of skin quality after fat grafting: clinical observation and an animal study. Plast Reconstr Surg. 2009 Sep;124(3):765-774. doi: 10.1097/PRS.0b013e3181b17b8f. PMID 19730294
- [Background] Khouri RK Jr, Khouri RE, Lujan-Hernandez JR, Khouri KR, Lancerotto L, Orgill DP. Diffusion and perfusion: the keys to fat grafting. Plast Reconstr Surg Glob Open. 2014 Oct 7;2(9):e220. doi: 10.1097/GOX.0000000000000183. eCollection 2014 Sep. PMID 25426403
- [Background] Tonnard P, Verpaele A, Peeters G, Hamdi M, Cornelissen M, Declercq H. Nanofat grafting: basic research and clinical applications. Plast Reconstr Surg. 2013 Oct;132(4):1017-1026. doi: 10.1097/PRS.0b013e31829fe1b0. PMID 23783059
- [Background] Xue EY, Narvaez L, Chu CK, Hanson SE. Fat Processing Techniques. Semin Plast Surg. 2020 Feb;34(1):11-16. doi: 10.1055/s-0039-3402052. Epub 2020 Feb 15. PMID 32071574
- [Background] Kling RE, Mehrara BJ, Pusic AL, Young VL, Hume KM, Crotty CA, Rubin JP. Trends in autologous fat grafting to the breast: a national survey of the american society of plastic surgeons. Plast Reconstr Surg. 2013 Jul;132(1):35-46. doi: 10.1097/PRS.0b013e318290fad1. PMID 23806907